CLINICAL TRIAL: NCT02939560
Title: Transcranial Magnetic Stimulation for Adults With Autism Spectrum Disorder and Depression
Brief Title: TMS for Adults With Autism and Depression
Acronym: TAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00056546
Record Dates: First submitted 2016-09-29; First posted 2016-10-20 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Autism Spectrum Disorder; Depression; Depressive Disorder; Major Depressive Disorder
Keywords: Autism Spectrum Disorder; Autism; Depressive; Depression
MeSH Terms: conditions — Autism Spectrum Disorder; Depression; Depressive Disorder; Depressive Disorder, Major; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rTMS (Experimental): Participants will receive rTMS sessions according to the study protocol.
  Interventions: Device: NeuroStar® TMS device (Neuronetics, Atlanta, GA)

INTERVENTIONS:
Device: NeuroStar® TMS device (Neuronetics, Atlanta, GA) — Participants in this study arm will be evaluated before and after receiving rTMS. Outcome measures will include social skills rating scales, depression rating scales and cognitive tasks while undergoing functional magnetic resonance imaging (fMRI).

SUMMARY:
The goal of this proposal is to investigate whether a standard rTMS protocol for depression, including multiple sessions applied to left dorsolateral prefrontal cortex (DLPFC) results in reduction of depressive symptoms for adult patients with ASD and MDD (Aim 1). The secondary goal is to investigate and whether there is any beneficial reduction in the core symptoms of autism (Aim 2).

DETAILED DESCRIPTION:
Aim 1. Determine the safety and therapeutic efficacy of left-sided DLPFC high frequency rTMS on MDD symptoms in patients with ASD: The investigators hypothesize that patients receiving the rTMS will tolerate the treatment course without difficulty and have clinically significant reduction of depressive symptoms after receiving all 25 sessions, as compared with their symptom burden prior to initiating TMS. Depression symptom data will be collected as pre- and post-TMS scores on Hamilton Depression Rating Scale (HAM-D). Depression scores will also be monitored periodically during course of TMS with Patient Health Questionnaires (PHQ-9).

Exploratory sub-aim - Monitoring for durability of response: The investigators hypothesize that subjects receiving rTMS will demonstrate durability of response in their depression symptom reduction, as measured by HAM-D scores at 1 month and 3 months post-TMS.

Aim 2. Determine the effect of left DLPFC rTMS on core symptoms of ASD: The investigators hypothesize that subjects will experience reduction in core symptoms of ASD after completing all 25 sessions, as compared with their symptom burden prior to initiating treatment. For social and communication deficits, informant and/or self-report evaluations will be made pre- and post-TMS with the Social Responsiveness Scale (SRS), the Ritvo Autism Aspergers Diagnostic Scale-Revised (RAADS-R) and the Aberrant Behavior Checklist (ABC). Repetitive and restricted behavior will be evaluated using the Repetitive Behavior Scale-Revised (RBS-R), the ABC, and RAADS.

Exploratory sub-aim: Determine if there are changes to functional brain connectivity during face and object processing tasks via functional MRI imaging in patients with Autism who receive rTMS: The study investigators hypothesize that there will be altered brain connectivity evident in patients' baseline fMRI during cognitive processing tasks prior to TMS reflected as both hyper- and hypo-connectivity, and that there will be some level of normalization of these patterns in fMRI after completion of TMS series, particularly in the prefrontal cortex.

Exploratory sub-aim - Monitoring for durability of response: The study investigators hypothesize that subjects receiving rTMS will exhibit durability of response in their ASD symptom reduction, as measured by ABC, SRS, RAADS, AND RBR scores at 1 month and 3 months post-TMS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autism Spectrum Disorder and active depressive symptoms.

Exclusion Criteria:

* List specific contraindicationsUncontrolled and/or untreated seizure disorder as defined by any incidence of seizure within the past 6 months. Patients with diagnosed epilepsy, or prior seizures, will be allowed in the study if they are taking an anticonvulsant medication, or have not had a seizure in the past year off medications.
* Moderate to severe intellectual disability (ID) as defined by IQ < 60, determined by prior IQ testing or Wechsler Abbreviated Scale of Intelligence (WASC-II) if no prior test results available
* Other psychiatric or neurodevelopmental illness that is the primary area of clinical focus (including but not limited to primary psychotic disorder, substance abuse disorder, and ASD or ID which are secondary to genetic syndromes)
* Active suicidal ideation or suicide attempt in the 90 days prior to initial assessment
* Presence of any metal implants or devices in the head or neck (e.g. metal plates or screws)
* No participants who are pregnant or who are planning to become pregnant
* Exclusion criteria for fMRI scanning:

  * have metal pins, plates or clips in the body or have orthodontics
  * have surgical implants such as pacemakers or cochlear implants
  * have permanent makeup or tattoos near the face or head
  * have metal fragments in the body (from welding, shrapnel, BB guns) or suspect that they have fragments
  * are claustrophobic
  * are pregnant
  * have ever suffered a closed head injury or concussion
  * are currently under the influence of alcohol or other recreational drugs
  * are a smoker
  * are currently enrolled in a course in which the PI or co-I's are instructors
  * cannot understand the task instructions
  * cannot lay still in the mock scanner for a period of 6 minutes
* Inability or unwillingness of participant or legal guardian/representative to give informed consent
* There will be no discrimination or exclusions based on race, gender, sexual orientation, or other socioeconomic factors. Of note, while both male and female participants will be actively and equally recruited using the same methods. The natural distribution of autism in the population skews towards significant towards male gender, with male prevalence being 4-5 times that of female prevalence. Our study will therefore likely have more male participants than female due to this trend in prevalence.
* Children (age <18) are being excluded from this study for several reasons. While autism is a pediatric neurodevelopmental disorder with symptom onset as young as one year of age, it is also one that is chronic throughout adulthood. Both children with autism and neurotypical children undergo periods of rapid change in brain size, structure, and organization as they age, and the interaction between a full rTMS series and brains that are still involved in periods of very active development and whom may also be at different points along their own developmental timelines may skew or alter the data that is collected. Additionally, due to both brain growth and increases in skull thickness, children of different ages may have significantly different "scalp to cortex" distances, which can result in very different patterns of cortical stimulation despite uniform coil positioning. This will be an added, unnecessary variable which would compromise the attempt at performing a standardized protocol. Finally, while high frequency rTMS is an FDA approved treatment for depression in adults, it has not yet been FDA approved in children and adolescents.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-09; Primary Completion 2018-06-01 (Actual); Study Completion 2018-09-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

REFERENCES:
- [Background] Perera T, George MS, Grammer G, Janicak PG, Pascual-Leone A, Wirecki TS. The Clinical TMS Society Consensus Review and Treatment Recommendations for TMS Therapy for Major Depressive Disorder. Brain Stimul. 2016 May-Jun;9(3):336-346. doi: 10.1016/j.brs.2016.03.010. Epub 2016 Mar 16. PMID 27090022
- [Background] Oberman LM, Enticott PG, Casanova MF, Rotenberg A, Pascual-Leone A, McCracken JT; TMS in ASD Consensus Group. Transcranial magnetic stimulation in autism spectrum disorder: Challenges, promise, and roadmap for future research. Autism Res. 2016 Feb;9(2):184-203. doi: 10.1002/aur.1567. Epub 2015 Nov 4. PMID 26536383
- [Result] George MS, Raman R, Benedek DM, Pelic CG, Grammer GG, Stokes KT, Schmidt M, Spiegel C, Dealmeida N, Beaver KL, Borckardt JJ, Sun X, Jain S, Stein MB. A two-site pilot randomized 3 day trial of high dose left prefrontal repetitive transcranial magnetic stimulation (rTMS) for suicidal inpatients. Brain Stimul. 2014 May-Jun;7(3):421-31. doi: 10.1016/j.brs.2014.03.006. Epub 2014 Mar 19. PMID 24731434
- [Result] Enticott PG, Fitzgibbon BM, Kennedy HA, Arnold SL, Elliot D, Peachey A, Zangen A, Fitzgerald PB. A double-blind, randomized trial of deep repetitive transcranial magnetic stimulation (rTMS) for autism spectrum disorder. Brain Stimul. 2014 Mar-Apr;7(2):206-11. doi: 10.1016/j.brs.2013.10.004. Epub 2013 Oct 27. PMID 24280031
- See also: Home page with information about the Primary Investigator — http://www.projectrex.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | rTMS
Started | 13
Completed | 10
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | rTMS
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 25.5 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hamilton Depression Rating Scale
Description: Hamilton Depression Rating Scale (HAM-D) with 17 questions. Minimum score = 0, maximum 53. Higher scores mean more severe depression.
Time Frame: Baseline through Week 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rTMS
Number analyzed (Participants) | 10
score on a scale
  Baseline | 21.5 (4.3)
  Week 5 | 10.2 (6.5)

2. Primary Outcome: Change From Baseline in Aberrant Behavior Checklist
Description: Aberrant Behavior Checklist. Minimum 0, maximum 174. Higher scores indicate worse behaviors.
Time Frame: Baseline, Week 5, Week 9, Week 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rTMS
Number analyzed (Participants) | 10
score on a scale
  Baseline | 53 (28)
  Week 5 | 24 (16)
  Week 9 | 20 (21)
  Week 17 | 30 (28)

3. Primary Outcome: Change From Baseline in Social Responsiveness Scale-2
Description: Social Responsiveness Scale-2. Minimum 0, maximum 195. Higher indicates worse behaviors
Time Frame: Baseline, Week 5, Week 9, Week 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rTMS
Number analyzed (Participants) | 10
score on a scale
  Baseline | 70.5 (10.6)
  Week 5 | 70.1 (14.3)
  Week 9 | 66.0 (16.6)
  Week 17 | 66.9 (15.0)

4. Primary Outcome: Change From Baseline in Ritvo Autism-Aspergers Diagnostic Scale
Description: Ritvo Autism-Aspergers Diagnostic Scale. Minimum 0, maximum 240. Higher indicates worse symptoms.
Time Frame: Baseline, Week 5, Week 9, Week 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rTMS
Number analyzed (Participants) | 10
score on a scale
  Baseline | 38 (11)
  Week 5 | 38 (15)
  Week 9 | 39 (14)
  Week 17 | 39 (15)

5. Primary Outcome: Change From Baseline in Repetitive Behavior Scale-Revised
Description: Repetitive Behavior Scale-Revised Global Impression. Minimum 0, maximum 100. Higher indicates worse behaviors
Time Frame: Baseline, Week 5, Week 9, Week 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | rTMS
Number analyzed (Participants) | 10
units on a scale
  Baseline | 59 (26)
  Week 5 | 26 (25)
  Week 9 | 27 (22)
  Week 17 | 30 (18)

6. Secondary Outcome: Change From Baseline in Functional MRI Scanning During Cognitive Processing Tasks
Description: Functional MRI data during cognitive processing tasks
Time Frame: Baseline, Week 5
Population: Unable to obtain due to lack of available equipment.
Arm/Group | rTMS
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline to 17 weeks
Arm/Group | rTMS
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 1/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rTMS (N=13)
Seizure (Nervous system disorders) | 1 (1) — Participant was administered brain stimulation outside of the safety range due to operator error.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/60/NCT02939560/Prot_SAP_000.pdf